CLINICAL TRIAL: NCT00002919
Title: PHASE II TRIAL OF THE COMBINATION OF TRANSURETHRAL RESECTION AND NEOADJUVANT CHEMOTHERAPY FOR PATIENTS WITH INVASIVE UROTHELIAL TRACT TUMORS SELECTED BY STAGE AND P53 NUCLEAR EXPRESSION
Brief Title: Combination Chemotherapy in Treating Patients With Stage II Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 96-066; CDR0000065305 (Registry Identifier: PDQ (Physician Data Query)); NCI-H97-1118
Record Dates: First submitted 1999-11-01; First posted 2004-03-12 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-07

CONDITIONS: Bladder Cancer
Keywords: stage II bladder cancer; transitional cell carcinoma of the bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Filgrastim; Cisplatin; Doxorubicin; Methotrexate; Vinblastine

INTERVENTIONS:
Biological: filgrastim
Drug: cisplatin
Drug: doxorubicin hydrochloride
Drug: methotrexate
Drug: vinblastine sulfate
Procedure: conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy following surgery in treating patients with stage II bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of combination chemotherapy with methotrexate, vinblastine, doxorubicin, and cisplatin (MVAC) following aggressive transurethral resection of bladder tumors in patients with stage II transitional cell carcinoma of the bladder without nuclear overexpression of mutant p53. II. Determine the proportion of patients treated with this regimen in whom bladder preservation rather than radical cystectomy is possible.

OUTLINE: All patients undergo complete or near complete transurethral resection of the bladder tumor at entry or within 6 weeks prior to entry. Upon confirmation of staging and histology, patients receive combination chemotherapy with methotrexate, vinblastine, doxorubicin, and cisplatin (MVAC) every 21 days for 4 courses. Subcutaneous G-CSF is given with each course. Patients with a complete response after chemotherapy proceed to intravesical therapy or observation; those with a partial response, stable disease, or progression proceed to definitive surgery.

PROJECTED ACCRUAL: 30 patients will be entered over approximately 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Invasive transitional cell carcinoma of the bladder that is clinical stage T2-3a N0 M0 by cystoscopy Cystoscopy performed at Memorial Sloan-Kettering Cancer Center (MSKCC) No multifocal carcinoma in situ No obstructive uropathy or palpable mass Pathologic confirmation of histology and no more than 20% positive expression of nuclear p53, as follows: On study following transurethral resection of the bladder (TURB) OR At TURB performed within 6 weeks of entry as part of initial staging

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60%-100% Hematopoietic: WBC at least 3,500 Platelets greater than 150,000 Hepatic: Bilirubin less than 2.0 mg/dL Renal: Creatinine less than 1.5 mg/dL OR Creatinine clearance greater than 60 mL/min per 1.73 square meters Cardiovascular: No NYHA class III/IV status Other: No concomitant malignancy other than basal cell skin carcinoma Negative pregnancy test required of fertile women Adequate contraception required of fertile women

PRIOR CONCURRENT THERAPY: No prior systemic chemotherapy No prior bladder irradiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 1996-11; Primary Completion 2003-01 (Actual); Study Completion 2003-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dean F. Bajorin, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States